CLINICAL TRIAL: NCT04046783
Title: Effectiveness and Tolerability of an Overnight 4-week Treatment With Patch Containing Onion Extract and Allantoin for Cesarean Section Scars
Brief Title: Patch With Onion Extract and Allantoin for C-section Scar
Status: Completed | Type: Observational
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Prof Valeria Conti, Professor, University of Salerno
Other Study IDs: USalerno
Record Dates: First submitted 2019-07-31; First posted 2019-08-06 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Cesarean Section; Dehiscence; Scar Keloid; Wound Heal
Keywords: Natural products; Wound healing; Cesarean delivery
MeSH Terms: conditions — Keloid | interventions — Transdermal Patch

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A included subjects without a history of C-section: Group A consisted of 47 women without a prior a history of C-section: 24 controls and 23 subjects who used patch. These latest 23 subjects applied overnight a patch containing a standardized quantity of Allium Cepa extract and allantoin on C-section scars over 4 weeks
  Interventions: Device: patch
- group B subjects who had already undergone previous C-section: Group B consisted of 46 women already undergone previous C-section: 22 controls and 24 subjects who used patch. These latest 24 subjects applied overnight a patch containing a standardized quantity of Allium Cepa extract and allantoin on C-section scars over 4 weeks
  Interventions: Device: patch

INTERVENTIONS:
Device: patch — an overnight application of a patch containing a standardized quantity of Allium Cepa extract and allantoin on C-section scars over 4 weeks.

SUMMARY:
The wound healing is a process occurring in response to dermal injury. The resulting scar may have various characteristics ranging from fine-line and asymptomatic to hypertrophic scars and keloids. Prevention or early treatment of pathological scars is the most appropriate approach. Among available remedies, gels and patches containing onion extract and allantoin have been demonstrated to be safe and effective in patients with scars of various origins and severity.

One of the most used natural products is a patch containing allium cepa and allantoin licensed for treatment of the scars including keloids. However, up to date, no controlled studies have evaluated the effects of such a device in women who have undergone Cesarean delivery. Therefore, the aim of this study was to investigate the effects of this patch on Cesarean section (C-section) scars.

DETAILED DESCRIPTION:
This is an observational non-interventional study. Women who underwent C-section were consecutively recruited at University Hospital of Salerno. Taking into account the number of C-section the study population was divided into two groups: Group A included subjects without a prior history of C-section, group B subjects who had already undergone previous C-section. At baseline after stitches removal, scars assessment was made using digital photographs and the validate Patient and Observer Scar Assessment Scale (POSAS). After 4 weeks, during the outpatient visit, women from both group A and B were asked whether had applied some natural products on the scars or not. In this occasion, the C-section of the women who had applied a patch containing allium cepa and allantoin as well as those of women who had not used any products (who represented the control group) were re-evaluated as at baseline. The Observers were blinded. One of them performed the scars assessment at baseline, the other one after 4 weeks. During the outpatient visit an informed consent for participation was obtained by all the subjects costituing the study population. The participation to the study was voluntary

ELIGIBILITY:
Inclusion Criteria:

* subjects undergone Cesarean delivery;
* age >18;
* voluntary participation to the study;
* informed consent release.

Exclusion Criteria:

* age <18
* hypersensitivity to any constituent of the patch;
* pre-term birth, obesity,
* gestational diabetes,
* hypertension,
* infections,
* dermatologic diseases
* use of both systemic and topic corticosteroids;
* no informed consent release.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women who have undergone Cesarean delivery
Study Population: The study population was represented by adult women, subdivided in two groups, A and B on the basis of the number of Cesearean delivery. Group A included subjects without a prior history of Cesarean delivery, Group B subjects who had already undergone previous Cesarean delivery. All the women were enrolled at University Hospital of Salerno, were >=18 years old without hypersensitivity to any constituent of the patch, who have not experienced pre-term birth, obesity, gestational diabetes, hypertension, infections, dermatologic diseases and use of both systemic and topic corticosteroids. All the partecipants were volunteers and released a written informed consent
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of an overnight 4-week Treatment with Patch containing Onion Extract and Allantoin for Cesarean Section Scars in women undergone to Cesarean section as assed by POSAS v.2.0. | Scars were evaluated at baseline and after 4 weeks by two observers and by the subjects.Scars assessment was made using digital photographs and the validate Patient and Observer Scar Assessment Scale (POSAS, version 2.0).
  The primary outcome was represented by the number of women undergone a Cesarean section (C-section) that used for 4-week a patch containing Allium Cepa extract and allantoin in respect to controls. The Patient and Observer Scar Assessment Scale (POSAS) was used to compare the differences from baseline to 4-week treatment and between controls and subjects using the patch

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Conti, PhD, Principal Investigator — Department of Medicine,University of Salerno, Baronissi (SA), Italy
Locations (1):
- University of Salerno, Dept. of Medicine, Baronissi, Campania, Italy

REFERENCES:
- [Result] Fearmonti RM, Bond JE, Erdmann D, Levin LS, Pizzo SV, Levinson H. The modified Patient and Observer Scar Assessment Scale: a novel approach to defining pathologic and nonpathologic scarring. Plast Reconstr Surg. 2011 Jan;127(1):242-247. doi: 10.1097/PRS.0b013e3181f959e8. PMID 21200219
- [Result] Gauglitz GG, Korting HC, Pavicic T, Ruzicka T, Jeschke MG. Hypertrophic scarring and keloids: pathomechanisms and current and emerging treatment strategies. Mol Med. 2011 Jan-Feb;17(1-2):113-25. doi: 10.2119/molmed.2009.00153. Epub 2010 Oct 5. PMID 20927486
- [Result] Prager W, Gauglitz GG. Effectiveness and Safety of an Overnight Patch Containing Allium cepa Extract and Allantoin for Post-Dermatologic Surgery Scars. Aesthetic Plast Surg. 2018 Aug;42(4):1144-1150. doi: 10.1007/s00266-018-1172-4. Epub 2018 Jun 14. PMID 29948103
- [Result] Willital GH, Heine H. Efficacy of Contractubex gel in the treatment of fresh scars after thoracic surgery in children and adolescents. Int J Clin Pharmacol Res. 1994;14(5-6):193-202. PMID 7672876
- [Result] Sidgwick GP, McGeorge D, Bayat A. A comprehensive evidence-based review on the role of topicals and dressings in the management of skin scarring. Arch Dermatol Res. 2015 Aug;307(6):461-77. doi: 10.1007/s00403-015-1572-0. Epub 2015 Jun 5. PMID 26044054
- [Result] Chuangsuwanich A, Jongjamfa K. The efficacy of combined herbal extracts gel preparation in the prevention of postsurgical hypertrophic scar formation. Dermatol Ther (Heidelb). 2014 Dec;4(2):187-95. doi: 10.1007/s13555-014-0055-0. Epub 2014 Jun 25. PMID 24962057
- [Result] Fang QQ, Chen CY, Zhang MX, Huang CL, Wang XW, Xu JH, Wu LH, Zhang LY, Tan WQ. The Effectiveness of Topical Anti-scarring Agents and a Novel Combined Process on Cutaneous Scar Management. Curr Pharm Des. 2017;23(15):2268-2275. doi: 10.2174/1381612822666161025144434. PMID 27784253
- [Result] Ho WS, Ying SY, Chan PC, Chan HH. Use of onion extract, heparin, allantoin gel in prevention of scarring in chinese patients having laser removal of tattoos: a prospective randomized controlled trial. Dermatol Surg. 2006 Jul;32(7):891-6. doi: 10.1111/j.1524-4725.2006.32192.x. PMID 16875470
- [Result] Rose P, Whiteman M, Moore PK, Zhu YZ. Bioactive S-alk(en)yl cysteine sulfoxide metabolites in the genus Allium: the chemistry of potential therapeutic agents. Nat Prod Rep. 2005 Jun;22(3):351-68. doi: 10.1039/b417639c. Epub 2005 May 10. PMID 16010345
- [Result] Pikula M, Zebrowska ME, Poblocka-Olech L, Krauze-Baranowska M, Sznitowska M, Trzonkowski P. Effect of enoxaparin and onion extract on human skin fibroblast cell line - therapeutic implications for the treatment of keloids. Pharm Biol. 2014 Feb;52(2):262-7. doi: 10.3109/13880209.2013.826246. Epub 2013 Sep 30. PMID 24074438
- [Result] Araujo LU, Grabe-Guimaraes A, Mosqueira VC, Carneiro CM, Silva-Barcellos NM. Profile of wound healing process induced by allantoin. Acta Cir Bras. 2010 Oct;25(5):460-6. doi: 10.1590/s0102-86502010000500014. PMID 20877959
- [Derived] Conti V, Corbi G, Iannaccone T, Corrado B, Giugliano L, Lembo S, Filippelli A, Guida M. Effectiveness and Tolerability of a Patch Containing Onion Extract and Allantoin for Cesarean Section Scars. Front Pharmacol. 2020 Sep 25;11:569514. doi: 10.3389/fphar.2020.569514. eCollection 2020. PMID 33101027